CLINICAL TRIAL: NCT02597673
Title: Trial of Self-managed Approaches for Patellofemoral Pain Syndrome in Active Duty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Blanchfield Army Community Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HU0001-15-1-TS08 (N15-P01)
Record Dates: First submitted 2015-10-05; First posted 2015-11-05 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2018-08

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard rehabilitation protocol (Active Comparator): Home Exercise Program (HEP). All participants will receive a standard home-based exercise rehabilitation protocol for PFPS. HEP teaches muscle strengthening exercises and self-management strategies to prevent recurrence. The HEP sessions provide the participant with a self-management framework for returning to duty following PFPS rehabilitation. The exercises are quadriceps strengthening exercises. These exercises consist of stretching exercises of the quadriceps and hamstring muscles and a combination of open chain and closed chain exercises. The combined open and closed chain exercises are active straight leg raises, quadriceps straightening, step up, and squats.
  Interventions: Other: Home Exercise Program (HEP)
- Self-Managed NMES Program (Experimental): Neuromuscular electrical stimulation (NMES). This group will receive a portable battery-operated device, KneeHAB® XP (Bio-Medical Research, Galway, Ireland) with the thigh garment. NMES training will consist of 20-minute stimulation sessions performed concurrently with the HEP for 9 weeks; each 20-minute NMES session includes a 2-minute warm-up, a 15-minute work-out and a 3-minute cool down. NMES with the thigh garment will be used as the participant is performing the home exercises of stretching and combined open and closed chain exercises. Those in the NMES group will alternate HEP alone and NMES with HEP for a total of 62 sessions (31 sessions of NMES/HEP and 31 sessions HEP alone).
  Interventions: Other: Home Exercise Program (HEP); Device: NMES
- Self-Managed TENS Program (Experimental): Transcutaneous electrical nerve stimulation (TENS). The TENS treatment groups will receive the battery-operated Kneehab® XP with lead wire TENS applicator system. The TENS protocol consists of 20-minutes of TENS stimulation while concurrently performing the HEP. The TENS with HEP and HEP alone will be alternated for 9 weeks for a total of 31 TENS/HEP sessions and 31 HEP alone for a total of 62 sessions.
  Interventions: Other: Home Exercise Program (HEP); Device: TENS
- Combined NMES/TENS Program (Experimental): The combined NMES/TENS treatment group will receive the Kneehab® XP with the conductive thigh garment and the lead wire TENS applicator. The same parameters for TENS and NMES will be used (described above). The NMES and the TENS protocol will be performed on alternating days. There will be a total of 31 NMES sessions with HEP and 31 TENS sessions with HEP for a total of 62 sessions.
  Interventions: Other: Home Exercise Program (HEP); Device: NMES; Device: TENS

INTERVENTIONS:
Other: Home Exercise Program (HEP) — All participants will receive a standard home-based exercise rehabilitation protocol for PFPS. HEP teaches muscle strengthening exercises and self-management strategies to prevent recurrence. This program includes sessions with the study coordinator. A handout and given a demonstration of the daily exercises to be performed at home and weekly communication from the study coordinator regarding compliance with the exercises.
Device: NMES — To ensure consistent interventions across participants, a specified percentage of baseline maximal voluntary contraction (% MVC) will be used to determine the intensity of the training contraction. The electrical amplitude to obtain the desired intensity will be determined for each participant. Participants will train at 20-30% of MVC during weeks 1-3, 30-40% of MVC during weeks 3-6, and 40-50% of MVC during weeks 6-9. Incremental increases will be made at the 3 and 6 week clinic visits. Individualized instructions for adjusting the amplitude dial settings, with a return demonstration, will be used to maintain the appropriate percentage of MVC. During the home training sessions, participants will adjust the amplitude required to achieve the desired goal, as tolerated.
  Other Names: KneeHAB® XP Thigh Garment
  Arms: Combined NMES/TENS Program; Self-Managed NMES Program
Device: TENS — The TENS protocol consists of 20-minutes of TENS stimulation while concurrently performing the HEP. The TENS with HEP and HEP alone will be alternated for 9 weeks. The Active device delivers a pre-set program of pulsed electrostimulation using a patented asymmetrical simple modulated pulse (SMP) waveform. SMP delivers a group of pulses as a repeating 12-second cycle.
  Other Names: KneeHAB® XP Lead Wire TENS Applicator
  Arms: Combined NMES/TENS Program; Self-Managed TENS Program

SUMMARY:
The overall objective of this project is to compare the three home-managed treatment regimens for PFPS: neuromuscular electrical stimulation (NMES), transcutaneous electrical nerve stimulation (TENS), and NMES combined with TENS to a standard home exercise program (HEP). Each of the three treatment arms will be supplemented by HEP and compared to a group receiving standard HEP alone. The central hypothesis is that the combination of NMES with TENS will show significantly greater improvements in muscle strength, mobility, pain, daily activity and quality of life (QOL) than HEP alone.

The investigators are examining: 1) whether the three treatment regimens are significantly more efficacious than standard HEP alone in improving lower extremity muscle strength, physical activity, mobility, pain, and quality of life; 2) lower extremity muscle strength, physical activity, mobility, pain, and quality of life differ significantly across the 4 time periods; 3) is there an interaction between treatment and time in relation to lower extremity muscle strength, physical activity, mobility, pain, and quality of life.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is the most common diagnosis among active duty military presenting with knee pain in the military ambulatory care setting. The incidence of PFPS has shown a striking increase of >11.3% over the last 4 years, affecting work performance, limiting activity, and impacting military deployment health. The investigators have shown that home-based neuromuscular electrical stimulation (NMES) is safe, portable, easy-to-use and improves quadriceps muscle strength with some pain relief. NMES and transcutaneous electrical nerve stimulation (TENS) devices are widely used by warfighters in the theatre of operation for knee problems. The overall objective of this project is to compare three home-managed treatment regimens for PFPS: NMES, TENS, and NMES combined with TENS to a standard home exercise program (HEP). The central hypothesis is that the combination of NMES with TENS will show significantly greater improvements in muscle strength, mobility, pain, daily activity and quality of life (QOL) than HEP alone. The rationale for this study is that increasing muscle strength and decreasing pain will significantly improve mobility, physical activity and QOL. Such outcomes will ultimately result in improved deployability, retention of military personnel and decreased economic costs in this population. The specific aims are to determine whether the three treatment regimens are significantly more efficacious than standard HEP for improving muscle strength, physical activity, mobility, QOL and symptoms of PFPS including pain. After consent and baseline testing, the investigators will randomly assign active duty male and female subjects, ages 18 to <45, (n=136) with PFPS to one of the four groups. Each of the three treatment arms will be supplemented by HEP and compared to a group receiving standard HEP alone. All groups will receive 9 weeks of home therapy. Using GEE methods, the investigators will build longitudinal regression models so that differences in time trends for the outcome variables among controls and those in the treatment groups can be statistically assessed. Positive results could translate into accelerated rehabilitation, decreased symptoms and lower medical costs with better patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

The study will be open to all active duty personal who are:

1. diagnosed with knee pain, categorized as anterior or retropatellar in one or both knees;
2. self-reported difficulty performing at least two or more of the following activities associated with knee pain: prolonged sitting, stair climbing, running, jumping and repetitive movements such as kneeling or squatting or stooping;
3. military service member at the time of diagnosis;
4. age ≥18 and <45 years; and
5. ability to provide freely given informed consent.

Exclusion Criteria:

Those who might be at risk of adverse outcomes from the study interventions will be excluded. This includes individuals with

1. Fracture or injury to external knee structures such that knee extension or flexion is impaired;
2. A significant co-morbid medical condition (such as severe hypertension, neurological disorder or pacemaker/defibrillator) in which NMES strength training or unsupervised exercise is contraindicated and would pose a safety threat or impair ability to participate;
3. Previous knee surgeries (i.e., tibiofemoral, patellofemoral) excluding knee arthroscopy;
4. Knee instability or recurrent patella dislocation or subluxation;
5. Inability or unwillingness to participate in a home exercise program or strengthening program;
6. Inability to speak and/or read English;
7. Reduced sensory perception in the lower extremities;
8. Pregnancy;
9. Vision impairment, where participant is classified as legally blind;
10. Unwillingness to accept random assignment; or
11. A score of 23 or greater on the Center for Epidemiological Studies-Depression scale (CES-D).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2015-07; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A Talbot, PhD EdD RN, Principal Investigator — University of Tennessee Health Sciences Center
Locations (1):
- Blanchfield Army Community Hospital, Fort Campbell North, Kentucky, United States

REFERENCES:
- [Background] The results of this study have not yet been published in a peer-reviewed journal. The registration will be updated with the full journal citation when the results are published.
- [Derived] Talbot LA, Solomon Z, Webb L, Morrell C, Metter EJ. Electrical Stimulation Therapies for Active Duty Military with Patellofemoral Pain Syndrome: A Randomized Trial. Mil Med. 2020 Aug 14;185(7-8):e963-e971. doi: 10.1093/milmed/usaa037. PMID 32248227

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants withdrew from the study during baseline testing, and prior to being assigned to a group.
Groups:
- Standard Rehabilitation Protocol: Home Exercise Program (HEP): HEP taught muscle strengthening exercises and self-management strategies. The exercises were quadriceps strengthening exercises that consist of stretching exercises of the quadriceps and hamstring muscles and a combination of open chain and closed chain exercises. The combined open and closed chain exercises were active straight leg raises, quadriceps straightening, step up, and squats.
- Self-Managed NMES Program: Neuromuscular electrical stimulation (NMES): NMES training consisted of 20-minute sessions performed concurrently with the HEP for 9 weeks; each 20-minute NMES session included a 2-minute warm-up, a 15-minute work-out and a 3-minute cool down. NMES with the thigh garment was used as the participant is performing the home exercises of stretching and combined open and closed chain exercises. Those in the NMES group received alternate HEP alone and NMES with HEP for a total of 62 sessions (31 sessions of NMES/HEP and 31 sessions HEP alone).
  Home Exercise Program (HEP): HEP taught muscle strengthening exercises and self-management strategies. The exercises were quadriceps strengthening exercises that consist of stretching exercises of the quadriceps and hamstring muscles and a combination of open chain and closed chain exercises. The combined open and closed chain exercises were active straight leg raises, quadriceps straightening, step up, and squats.
- Self-Managed TENS Program: Transcutaneous electrical nerve stimulation (TENS). The TENS treatment groups received the battery-operated Kneehab® XP with lead wire TENS applicator system. The TENS protocol consisted of 20-minutes of TENS stimulation while concurrently performing the HEP. The TENS with HEP and HEP alone was alternated for 9 weeks for a total of 31 TENS/HEP sessions and 31 HEP alone for a total of 62 sessions.
  Home Exercise Program (HEP): HEP taught muscle strengthening exercises and self-management strategies. The exercises were quadriceps strengthening exercises that consist of stretching exercises of the quadriceps and hamstring muscles and a combination of open chain and closed chain exercises. The combined open and closed chain exercises were active straight leg raises, quadriceps straightening, step up, and squats.
- Combined NMES/TENS Program: The combined NMES/TENS treatment group received the Kneehab® XP with the conductive thigh garment and the lead wire TENS applicator. The same parameters for TENS and NMES were used (described above). The NMES and the TENS protocol were performed on alternating days. There was a total of 31 NMES sessions with HEP and 31 TENS sessions with HEP for a total of 62 sessions.
  Home Exercise Program (HEP): HEP taught muscle strengthening exercises and self-management strategies. The exercises were quadriceps strengthening exercises that consist of stretching exercises of the quadriceps and hamstring muscles and a combination of open chain and closed chain exercises. The combined open and closed chain exercises were active straight leg raises, quadriceps straightening, step up, and squats.
Period: Overall Study
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Started | 34 | 33 | 33 | 30
Completed | 31 | 27 | 28 | 25
Not Completed | 3 | 6 | 5 | 5

BASELINE CHARACTERISTICS:
Population: Talbot LA, Soloman Z, Webb L, Morrell C, Metter EJ. (In Press) Electrical Stimulation Therapies for Active Duty Military with Patellofemoral Pain Syndrome: A Randomized Trial. Military Medicine. Manuscript number: MILMED-D-19-00678.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program | Total
Number analyzed (Participants) | 34 | 33 | 33 | 30 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 34 | 33 | 33 | 30 | 130
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 6 | 29
  Male | 26 | 25 | 26 | 24 | 101
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 2 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 5 | 11 | 13 | 41
  White | 17 | 21 | 15 | 17 | 70
  More than one race | 3 | 5 | 4 | 0 | 12
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 33 | 30 | 130
Height [Mean (Standard Deviation); unit: cm] | 176 (11.2) | 174 (10.8) | 177 (8.1) | 175 (7.37) | 176 (9.5)
Weight [Mean (Standard Deviation); unit: kg] | 86 (16.7) | 85 (16.1) | 86 (14.4) | 84 (14.8) | 85.3 (15.4)

OUTCOME MEASURES:

1. Primary Outcome: Lower Extremity Muscle Strength- Extension
Description: The NMMT is a handheld device which measures knee extensor (KE) and flexor (KF) muscle strength. The measurement of KE strength on the PFPS leg is reported. For each test, participants performed three maximal efforts holding each contraction for 4 seconds, separated by 30-second rest; the highest value of the three trials will be accepted in kilograms.
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: Kg-Force
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Number analyzed (Participants) | 34 | 33 | 33 | 30
Kg-Force
  Injured Knee: Week 0 | 41.58 (16.56) | 37.74 (15.39) | 37.14 (15.36) | 40.42 (18.87)
  Injured Knee: Week 3 | 41.41 (14.92) | 42.70 (18.66) | 43.21 (21.49) | 43.07 (17.80)
  Injured Knee: Week 6 | 44.35 (12.40) | 43.31 (17.52) | 41.67 (20.60) | 43.03 (16.54)
  Injured Knee: Week 9 | 41.78 (13.46) | 46.22 (18.31) | 45.44 (23.16) | 46.89 (17.78)
  Unaffected Knee: Week 0 | 45.07 (17.83) | 44.56 (18.75) | 43.75 (17.33) | 45.42 (18.67)
  Unaffected Knee: Week 3 | 42.81 (15.79) | 47.16 (19.24) | 46.64 (18.58) | 44.61 (18.60)
  Unaffected Knee: Week 6 | 42.74 (14.50) | 47.58 (18.51) | 46.31 (16.60) | 46.14 (15.84)
  Unaffected Knee: Week 9 | 43.83 (14.72) | 47.87 (20.64) | 46.69 (18.93) | 50.62 (18.32)

2. Primary Outcome: Lower Extremity Muscle Strength- Flexion
Description: as for outcome 1
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: Kg-Force
Groups:
- Self-Managed TENS Program: Transcutaneous electrical nerve stimulation (TENS). The TENS treatment groups received the battery-operated Kneehab® XP with lead wire TENS applicator system. The TENS protocol consisted of 20-minutes of TENS stimulation while concurrently performing the HEP. The TENS with HEP and HEP alone was alternated for 9 weeks for a total of 31 TENS/HEP sessions and 31 HEP alone for a total of 62 sessions.
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Number analyzed (Participants) | 34 | 33 | 33 | 30
Kg-Force
  Injured Knee: Week 0 | 21.85 (7.61) | 20.32 (7.35) | 21.33 (7.13) | 21.95 (9.13)
  Injured Knee: Week 3 | 22.07 (8.05) | 22.49 (8.76) | 22.99 (8.04) | 22.56 (8.84)
  Injured Knee: Week 6 | 22.84 (7.36) | 23.72 (7.35) | 22.43 (8.76) | 23.86 (8.47)
  Injured Knee: Week 9 | 24.15 (9.67) | 26.95 (8.17) | 25.01 (9.11) | 26.64 (10.02)
  Unaffected Knee: Week 0 | 23.89 (7.20) | 23.11 (7.30) | 24.34 (7.50) | 25.20 (8.67)
  Unaffected Knee: Week 3 | 24.71 (8.58) | 24.93 (8.49) | 23.93 (7.95) | 24.40 (8.43)
  Unaffected Knee: Week 6 | 25.13 (8.80) | 24.64 (7.53) | 23.65 (8.61) | 25.20 (7.79)
  Unaffected Knee: Week 9 | 24.54 (8.27) | 26.21 (8.16) | 25.30 (8.30) | 26.96 (8.53)

3. Primary Outcome: Lower Extremity Strength- 30-Second Chair Stand Test
Description: Mobility was measured by the number of complete standing and sitting cycles in 30-seconds
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: rises
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Number analyzed (Participants) | 34 | 33 | 33 | 30
rises
  Week 0 | 11.6 (2.8) | 11.0 (3.0) | 11.0 (3.1) | 11.0 (3.8)
  Week 3 | 13.2 (3.5) | 12.3 (4.0) | 11.7 (3.0) | 12.6 (4.1)
  Week 6 | 14.2 (3.4) | 12.8 (4.4) | 13.0 (2.9) | 13.6 (3.9)
  Week 9 | 15.3 (4.0) | 14.4 (4.4) | 13.4 (3.5) | 15.1 (4.8)

4. Primary Outcome: Lower Extremity Strength- Timed Stair Climb Test
Description: Strength, balance, and power were measured by the number seconds it took to ascend and descend 4 steps (6 in rise, 11.5 in run).
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Number analyzed (Participants) | 34 | 33 | 33 | 30
Seconds
  Week 0 | 3.7 (1.1) | 4.0 (1.4) | 4.2 (1.4) | 4.1 (1.6)
  Week 3 | 3.6 (0.8) | 3.7 (1.0) | 3.8 (1.0) | 3.6 (1.3)
  Week 6 | 3.4 (0.6) | 3.5 (1.1) | 3.7 (0.9) | 3.7 (0.9)
  Week 9 | 3.3 (0.7) | 3.5 (1.2) | 3.3 (1.0) | 3.4 (0.9)

5. Primary Outcome: Lower Extremity Mobility- Forward Step-down Test
Description: Mobility was measured by the number of step down repetitions completed in 30 seconds.
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: Number of Repetitions
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Number analyzed (Participants) | 34 | 33 | 33 | 30
Number of Repetitions
  Week 0 | 13.2 (3.9) | 11.3 (3.6) | 10.8 (4.9) | 11.2 (4.0)
  Week 3 | 15.4 (5.0) | 12.9 (4.3) | 11.8 (4.8) | 14.4 (5.6)
  Week 6 | 17.0 (4.9) | 14.0 (5.6) | 13.9 (5.4) | 15.3 (4.9)
  Week 9 | 17.7 (5.2) | 16.3 (5.3) | 14.9 (5.7) | 18.0 (6.0)

6. Primary Outcome: Lower Extremity Mobility- 6-Minute Walk Test
Description: Mobility was measured by the distance walked at a fast pace over 6-minutes.
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: Inches
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Number analyzed (Participants) | 34 | 33 | 33 | 30
Inches
  Week 0 | 24612 (2964) | 23931 (2772) | 23999 (2979) | 23174 (2638)
  Week 3 | 24373 (3053) | 24919 (2804) | 24951 (3407) | 24102 (2996)
  Week 6 | 24970 (2582) | 25772 (3204) | 25284 (3426) | 24753 (2311)
  Week 9 | 25059 (3073) | 25892 (3300) | 25847 (3763) | 25227 (2655)

7. Secondary Outcome: Current Knee Pain
Description: Current Knee Pain was assessed using the Visual Analog Scale, an 11-point numerical rating scale. Participants rated current knee pain intensity on a scale of 0 (no pain) to 10 (worst pain imaginable). A mean pain score was calculated.
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Number analyzed (Participants) | 34 | 33 | 33 | 30
score on a scale
  Week 0 | 3.48 (1.84) | 3.42 (1.66) | 4.24 (1.76) | 3.98 (1.77)
  Week 3 | 2.99 (1.99) | 2.78 (1.71) | 3.44 (2.13) | 3.02 (1.91)
  Week 6 | 2.90 (2.20) | 2.28 (1.50) | 3.76 (2.05) | 2.72 (1.80)
  Week 9 | 2.77 (2.22) | 2.44 (1.79) | 3.01 (2.33) | 3.27 (2.26)

8. Secondary Outcome: Knee Pain Following Performance Testing- 30-Second Chair Stand Test
Description: Knee pain intensity after the 30-Second Chair Stand Test was assessed using the Visual Analog Scale, an 11-point numerical rating scale. Participants rated current knee pain intensity on a scale of 0 (no pain) to 10 (worst pain imaginable). A mean pain score was calculated.
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Number analyzed (Participants) | 34 | 33 | 33 | 30
score on a scale
  Week 0 | 2.9 (1.8) | 2.8 (1.7) | 3.9 (1.8) | 3.6 (2.0)
  Week 3 | 2.9 (1.9) | 2.2 (1.7) | 3.5 (2.0) | 2.9 (2.2)
  Week 6 | 2.8 (2.2) | 2.3 (1.7) | 3.6 (2.1) | 2.9 (2.3)
  Week 9 | 2.8 (2.2) | 2.5 (1.9) | 2.6 (2.2) | 2.6 (2.4)

9. Secondary Outcome: Knee Pain Following Performance Testing- Stair Climb Test
Description: Knee pain intensity after the Stair Climb Test was assessed using the Visual Analog Scale, an 11-point numerical rating scale. Participants rated current knee pain intensity on a scale of 0 (no pain) to 10 (worst pain imaginable). A mean pain score was calculated.
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Number analyzed (Participants) | 34 | 33 | 33 | 30
score on a scale
  Week 0 | 2.7 (1.9) | 2.7 (1.8) | 3.5 (1.9) | 3.0 (2.2)
  Week 3 | 2.6 (2.1) | 2.3 (1.5) | 3.4 (2.0) | 2.4 (2.1)
  Week 6 | 2.7 (2.0) | 2.1 (1.7) | 3.6 (2.3) | 2.2 (2.1)
  Week 9 | 2.7 (2.0) | 2.0 (1.8) | 2.7 (2.3) | 1.9 (2.1)

10. Secondary Outcome: Knee Pain Following Performance Testing- Forward Step Down Test
Description: Knee pain intensity after the Forward Step Down Test was assessed using the Visual Analog Scale, an 11-point numerical rating scale. Participants rated current knee pain intensity on a scale of 0 (no pain) to 10 (worst pain imaginable). A mean pain score was calculated.
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Number analyzed (Participants) | 34 | 33 | 33 | 30
score on a scale
  Week 0 | 4.2 (1.5) | 4.2 (2.2) | 5.2 (1.9) | 5.3 (2.1)
  Week 3 | 3.8 (2.0) | 3.2 (2.0) | 4.7 (2.0) | 3.5 (2.3)
  Week 6 | 3.6 (2.2) | 3.3 (1.7) | 4.2 (2.1) | 3.6 (2.2)
  Week 9 | 3.5 (2.2) | 2.8 (2.1) | 3.3 (2.1) | 3.2 (2.5)

11. Secondary Outcome: Knee Pain Following Performance Testing- 6-Minute Walk Test
Description: Knee pain intensity after the 6-Minute Walk Test was assessed using the Visual Analog Scale, an 11-point numerical rating scale. Participants rated current knee pain intensity on a scale of 0 (no pain) to 10 (worst pain imaginable). A mean pain score was calculated.
Time Frame: 0, 3, 6, and 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
Number analyzed (Participants) | 34 | 33 | 33 | 30
score on a scale
  Week 0 | 3.2 (1.7) | 2.7 (2.2) | 4.5 (1.7) | 3.6 (2.3)
  Week 3 | 3.3 (2.0) | 2.5 (1.6) | 4.3 (2.0) | 3.2 (2.2)
  Week 6 | 3.1 (2.2) | 2.9 (2.1) | 3.9 (2.4) | 2.6 (1.9)
  Week 9 | 3.0 (2.1) | 2.3 (2.0) | 2.9 (2.3) | 2.7 (2.5)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Standard Rehabilitation Protocol | Self-Managed NMES Program | Self-Managed TENS Program | Combined NMES/TENS Program
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 0/33 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/33 | 0/30
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/33 | 0/30

LIMITATIONS AND CAVEATS:
Refer to: TalbotLA, SolomanZ, WebbL, MorrellC, MetterEJ.(2020)Electrical Stimulation Therapies for Active Duty Military with Patellofemoral Pain Syndrome:A Randomized Trial. Mil Med 2020Apr6 pii:usaa037 doi:10.1093/milmed/usaa037[Epub ahead of print]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT02597673/Prot_000.pdf
  • Statistical Analysis Plan (2015-07-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT02597673/SAP_001.pdf